CLINICAL TRIAL: NCT02010411
Title: Effects of Prolastin Aerosol Therapy on Bacterial Density in the Airways of Patients With Cystic Fibrosis
Brief Title: Alpha1 Antitrypsin Aerosol Therapy in Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Technical problems with measure of CFU's. Outcomes published: PMID:16986483
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Cantin, Doctor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-038
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — alpha 1-Antitrypsin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prolastin (Active Comparator): Prolastin 250 mg nebulized BID, 10 days
  Interventions: Drug: Prolastin (drug)

INTERVENTIONS:
Drug: Prolastin (drug) — Outcomes compared to saline or no intervention in each subject.
  Other Names: Alpha1 antitrypsin

SUMMARY:
The hypothesis being tested is that inhibition of the enzyme known as elastase in the airways of patients with cystic fibrosis will help decrease the number of bacteria. Alpha1 antitrypsin, an elastase inhibitor, will be given to patients with cystic fibrosis by aerosol therapy twice in 1 day and sputum will be collected to measure the density of bacteria

DETAILED DESCRIPTION:
Cystic fibrosis is usually characterized by chronic bacterial infections of the airways. Neutrophils release the enzyme elastase in the airways and this enzyme can prevent the ingestion and killing of bacteria by the airway phagocytic cells. The hypothesis being tested is that inhibition of elastase in the airways will help neutrophils decrease the number of bacteria. Each subject with cystic fibrosis will first undergo aerosol therapy with a sterile saline solution and sputum will be collected 2, 4 and 6 hours after the aerosol therapy to measure the density of bacteria. Subsequently, alpha1 antitrypsin, an elastase inhibitor, will be given to the same patients by aerosol therapy twice in 1 day and sputum will be collected at 2, 4 and 6 hours after treatment to measure the density of bacteria. The results will be compared to those obtained after after aerosol therapy with saline solution.

Study phase II

Study type Interventional

Study design Purpose - treatment Allocation - nonrandomized trial Masking - open Control - active Assignment - cross-over Endpoint - efficacy

Primary Outcome Measure Bacterial density in sputum as determined by colony forming units at 2, 4 and 6 hours after Prolastin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Age 14 years and older
* Women must have a negative pregnancy test and used effective contraception
* Must be able to produce sputum
* Sputum culture positive for Pseudomonas aeruginosa

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-06; Primary Completion 2004-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bacterial density in sputum as determined by colony forming units at 2, 4 and 6 hours after Prolastin therapy. | 6 hours after Prolastin

SECONDARY OUTCOMES:
Neutrophil burden in airways as determined by sputum myeloperoxidase; | 6 hours after Prolastin
Sputum elastase activity | 6 hours after Prolastin
Alpha1 antitrypsin in sputum | 6 hours after Prolastin

CONTACTS AND LOCATIONS:
Overall Officials: Andre Cantin, md, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] McElvaney NG, Hubbard RC, Birrer P, Chernick MS, Caplan DB, Frank MM, Crystal RG. Aerosol alpha 1-antitrypsin treatment for cystic fibrosis. Lancet. 1991 Feb 16;337(8738):392-4. doi: 10.1016/0140-6736(91)91167-s. PMID 1671425